CLINICAL TRIAL: NCT00206700
Title: Open-label Trial of Leukine® (Sargramostim), A Recombinant Human Granulocyte-Macrophage Colony Stimulating Factor (GM-CSF), in Active Crohn's Disease
Brief Title: Open-label Trial of Leukine in Active Crohn's Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 307340; 91274; Novel 5; NCT00185471 (obsolete NCT alias)
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-12

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — sargramostim

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Sargramostim (Leukine)

INTERVENTIONS:
Drug: Sargramostim (Leukine) — Open Label, 8 week cycle
  Other Names: BAY86-5326

SUMMARY:
The purpose of this study is to establish a safety profile sargramostim administered in 8 week cycles to adult patients with active Crohn's disease.

DETAILED DESCRIPTION:
On 29 May 2009, Bayer began transitioning the sponsorship of this trial to Genzyme. NOTE: This study was originally posted by sponsor Berlex, Inc. Berlex, Inc. was renamed to Bayer HealthCare, Inc.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent
* Participated in a previous study of sargramostim in Crohn's disease within the past 12 months
* Subjects who participated in protocols excluding concomitant steroid use:
* Must have moderately to severely active Crohn's disease at time of screening (CDAI score >/= 220 points and less than or equal to 475 points)
* Must be receiving less than or equal to 40 mg prednisone (or equivalent) daily at time of screening if treated with corticosteroids between completing their previous sargramostim study and entry into this study and be able to taper to less than or equal to 7.5 mg daily within one treatment cycle
* Subjects who participated in Protocol 307501
* Must have active Crohn's disease (CDAI score > 150 points and less than or equal to 450 points) if completely withdrawn from CS use
* Must be receiving less than or equal to 40 mg prednisone (or equivalent) daily at time of screening, be able to taper to less than or equal to 7.5 mg daily within 2 treatment cycles, and have a CDAI score less than or equal to 450 points if not completely withdrawn from CS use
* Have a negative serum pregnancy test within 2 weeks prior to receiving initial dose of sargramostim in female subjects of child-bearing potential (optional - may be waived by the investigator if the subject has had no interruption in contraception method since participation in the previous study)
* Agree to use of an adequate method of contraception throughout the study period for sexually-active males and females of childbearing potential
* Able to self-inject sargramostim or have a designee who can do so
* Able to comply with protocol requirements
* Have a negative stool exam if subject received a course of antibiotics since participation in the previous study

Exclusion Criteria:

* Pregnant or breastfeeding female
* Need for gastrointestinal (GI) surgery for active GI bleeding, peritonitis, intestinal obstruction, or intra-abdominal or perianal abscess requiring surgical drainage
* Gastrointestinal surgery within the prior 6 months
* Symptoms of bowel obstruction or confirmed evidence of a clinically-significant stricture within the last 6 months that has not been surgically corrected
* Serum creatinine greater than or equal to 2.0 mg/dL
* Alkaline phosphatase (ALP), aspartate aminotransferase (AST), alanine aminotransferase (ALT), or total bilirubin greater or equal to 2X the upper limit of normal; hemoglobin (Hb) < 8.0 gm/dL; platelet count greater than or equal to 800,000/mL; ANC less than or equal to 1,000/µL or > 20,000/µL (the exclusion of subjects with ANC > 20,000/µL applies only to entry into the first treatment cycle)
* Use of licensed/registered anti-tumor necrosis factor (TNF) therapy such as infliximab within 8 weeks prior to first dose of study drug in this trial
* Use of any of the following medications within 4 weeks prior to receiving the first dose of study drug: 6-mercaptopurine, azathioprine, cyclophosphamide, methotrexate, mycophenolate mofetil, tacrolimus, cyclosporine, or thalidomide
* Use of any experimental agent in a clinical trial since participating in a sargramostim trial
* History of allergy to yeast products or sargramostim
* Psychiatric illness or substance abuse that would interfere with ability to comply with protocol requirements or give informed consent
* Clinically important primary disease unrelated to Crohn's disease
* Prior exposure to natalizumab (Tysabri)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 378 (Actual)
Dates: Start 2003-02; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
To establish a safety profile for long-term, repeated cycles of sargramostim administered to subjects with Crohn's disease. | Not applicable for this outcome

SECONDARY OUTCOMES:
Crohn's disease activity | After successive 8-week cycles of treatment
Duration of clinical remission and time to disease flare | After successive cycles of sargramostim therapy
Patient compliance | After successive cycles of sargramostim therapy

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (141):
- United States (83):
  - Birmingham, Alabama
  - Scottsdale, Arizona
  - Berkeley, California
  - Los Angeles, California
  - Orange, California
  - San Francisco, California
  - Tarzana, California
  - Aurora, Colorado
  - Englewood, Colorado
  - Lakewood, Colorado
  - Littleton, Colorado
  - Washington D.C., District of Columbia
  - Boca Raton, Florida
  - Clearwater, Florida
  - Gainesville, Florida
  - Hollywood, Florida
  - Jacksonville, Florida
  - North Miami Beach, Florida
  - Winter Park, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Lake Charles, Louisiana
  - Metairie, Louisiana
  - Slidell, Louisiana
  - Annapolis, Maryland
  - Hagerstown, Maryland
  - Towson, Maryland
  - Boston, Massachusetts
  - Chesterfield, Michigan
  - Troy, Michigan
  - Plymouth, Minnesota
  - Mexico, Missouri
  - St Louis, Missouri
  - Billings, Montana
  - Lincoln, Nebraska
  - Lebanon, New Hampshire
  - Berlin, New Jersey
  - Great Neck, New York
  - Mineola, New York
  - New York, New York
  - Rochester, New York
  - Syracuse, New York
  - Asheville, North Carolina
  - Chapel Hill, North Carolina
  - Charlotte, North Carolina
  - Greensboro, North Carolina
  - Wilmington, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Portland, Oregon
  - Hanover, Pennsylvania
  - Lancaster, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Sayre, Pennsylvania
  - Charleston, South Carolina
  - Columbia, South Carolina
  - Bristol, Tennessee
  - Jackson, Tennessee
  - Kingsport, Tennessee
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Dallas, Texas
  - Irving, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Charlottesville, Virginia
  - Chesapeake, Virginia
  - Danville, Virginia
  - Norfolk, Virginia
  - Richmond, Virginia
  - Bellevue, Washington
  - Seattle, Washington
  - Spokane, Washington
  - Walla Walla, Washington
  - Wenatchee, Washington
  - Madison, Wisconsin
  - Milwaukee, Wisconsin
- Buenos Aires, Buenos Aires F.D., Argentina
- Australia (14):
  - Garran, Australian Capital Territory
  - Concord, New South Wales
  - New Lambton Heights, New South Wales
  - Sydney, New South Wales
  - Brisbane, Queensland
  - Adelaide, South Australia
  - Launceston, Tasmania
  - Ballarat, Victoria
  - Frankston, Victoria
  - Melbourne, Victoria
  - Parkville, Victoria
  - Prahran, Victoria
  - Fremantle, Western Australia
  - Penrith
- Brazil (5):
  - Salvador, Estado de Bahia
  - Curitiba, Paraná
  - Rio de Janeiro, Rio de Janeiro
  - Porto Alegre, Rio Grande do Sul
  - São Paulo, São Paulo
- Canada (10):
  - Edmonton, Alberta
  - Kelowna, British Columbia
  - Vancouver, British Columbia
  - Winnipeg, Manitoba
  - Hamilton, Ontario
  - London, Ontario
  - Toronto, Ontario
  - Windsor, Ontario
  - Montreal, Quebec
  - Québec, Quebec
- New Zealand (4):
  - Milford, Auckland
  - Auckland
  - Christchurch
  - Hamilton
- Russia (6):
  - Lipetsk, Russia
  - Moskva, Russia
  - Samara, Russia
  - Moscow
  - Moskva
  - Volgograd
- Switzerland (3):
  - Basel, Basel
  - Bern, Canton of Bern
  - Lausanne, Canton of Vaud
- Ukraine (5):
  - Donetsk
  - Kharkiv
  - Kiev
  - Lviv
  - Vinnitsa
- United Kingdom (10):
  - Bristol, Avon
  - London, Greater London
  - Salford, Greater Manchester
  - Edinburgh, Lothian
  - Liverpool, Merseyside
  - Harrow, Middlesex
  - Cardiff, South Glamorgan
  - Newcastle upon Tyne, Tyne and Wear
  - London
  - Sheffield